CLINICAL TRIAL: NCT02261779
Title: Phase I/II Pilot Trial of ATRA (Tretinoin) and TCP (Tranylcypromine) in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) and no Intensive Treatment is Possible
Brief Title: Phase I/II Trial of ATRA and TCP in Patients With Relapsed or Refractory AML and no Intensive Treatment is Possible
Acronym: TCP-AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Dr. Petra Tschanter, Dr.med.Petra Tschanter, Martin-Luther-Universität Halle-Wittenberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM_04_12_TCP_ATRA_AML; 2012-002154-23 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-10-10 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: AML
MeSH Terms: interventions — Tranylcypromine; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tretinoin & Tranylcypromine (Experimental): Tretinoin started with 45mg/m2 on day 7 for one year, administered orally as soft capsules, Tranylcypromine started with 10mg/d up to a maximum dose of 60mg/d for on year, administered orally as tablets
  Interventions: Drug: Tranylcypromine; Drug: Tretinoin

INTERVENTIONS:
Drug: Tranylcypromine
  Other Names: Jatrosom
Drug: Tretinoin
  Other Names: Vesanoid

SUMMARY:
Longterm disease-free survival (DFS) of older patients with acute myeloid leukemia (AML) remains poor. The vast majority of AML patients relapses within two years after start of therapy1,2. In Acute Promyelocytic Leukemia (APL, AML M3), all-trans-retinoic-acid (ATRA; Tretinoin) induces differentiation and subsequently clinical remission. So far effective differentiation therapy does not exist in other AML subtypes. Recent preclinical data suggest that the combinatorial use of ATRA and tranylcypromine (TCP), an irreversible Monoamine-Oxidase (MAO) and Lysin-specific demethylase (LSD) inhibitor that also inhibits LSD1 (a histone H3 Lysine 4 demethylase), induces leukemia cell differentiation and leukemic stem cell exhaustion in vitro and in vivo in non-APL AML subtypes.

In this Phase I/II study the investigators will explore the feasibility, safety, as well as efficacy and of Tretinoin/TCP treatment in patients with relapsed or refractory AML or in patients with AML who are not eligible for intensive treatment. Patients will be treated with daily increasing doses of TCP (initially 10 mg/day, then +10 mg each day up to 80mg/d). After 7 days, ATRA will be added at a fixed dose (45 mg/sqm/day). Overall, 16 evaluable patients are going to be treated. The primary endpoint is the fraction of patients that achieve CR, CRp( complete response with incomplete recovery of platelets), CRi (complete response with incomplete recovery of granulocytes) and PR. Secondary endpoints are tolerability, safety as well as progression-free survival and overall survival. Serum levels of TCP will be regularly analyzed. Pharmacodynamic analyses will be performed with analyses of the inhibition of LSD1 by TCP. Further analyses will address the changes in Histone H3 lysine 4 tri demethylase (H3K4me3) levels in AML blasts and the differentiation status of AML blasts.

Taken together, this Phase I/II study will analyze feasibility, pharmacodynamics and effectivity of ATRA and TCP as differentiation therapy in AML.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments which are not routinely performed for diagnosis or monitoring of AML, and the subjects must be willing to comply with treatment and to follow up assessments and procedures
2. Histologically or cytologically confirmed diagnosis of AML relapsed after or refractory to at least one induction regimen, or patients with AML at initial diagnosis who are not eligible for allogeneic transplant or intensive induction chemotherapy (investigator´s choice; for example reduced general state), except for AML M3 (acute promyelocytic leukemia).
3. Age > 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤3 (see Appendix, 3.2)
5. Measurable disease burden (blasts in bonemarrow (BM) and/or peripheral blood (PB), extramedullary blasts [chloroma])
6. Able to swallow and retain oral medication
7. A life expectancy of at least 4 weeks
8. Adequate contraception methods
9. Adequate organ function

Exclusion Criteria:

1. Patients with more than 20.000/µl leukocytes in the peripheral blood that cannot be controlled by Hydroxyurea.
2. Patients with a valid option for intensive chemotherapy and/ or stem cell transplantation. (Patients after allogeneic stem cell transplant must be off immunosuppressive agents for at least 2 weeks prior to study entry and Graft- versus host disease must have resolved to Grade <= 2)
3. Patients with less than 30% blasts in the bone marrow at the time of diagnosis. They should receive Azacytidine monotherapy.
4. History of cancer that according to the Investigator might confound the assessment of the endpoints of the study
5. Uncontrolled peptic ulcer disease or clinically significant gastrointestinal abnormalities which interfere with oral dosing or any unstable or serious concurrent condition (e.g., active uncontrolled infection)
6. Poorly controlled hypertension (defined as systolic blood pressure (SBP) of ≥170 mmHg). Note: Initiation or adjustment of antihypertensive medication is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/ DBP(diastolic blood pressure) values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for he study.
7. Prolongation of corrected QT interval (QTc) > 480 ms
8. History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction (MI), unstable angina, symptomatic peripheral vascular disease, class 3 or 4 congestive heart failure, as defined by the New York Heart Association (NYHA)
9. Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
10. History of cerebrovascular infarction or bleeding, pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti- coagulant agents for at least 6 weeks are eligible
11. Evidence of serious active bleeding or bleeding diathesis (except for bleeding or petechiae due to AML- related thrombocytopenia which will be treated using platelet transfusions). Also, patients with known endobronchial lesions and/ or lesions infiltrating major pulmonary vessels will be excluded from the study due to excess risk of bleeding.
12. Prior major surgery or trauma within 28 days prior to first dose of study drug
13. Treatment with an investigational agent within 21 days or 5 half-life, whichever is longer prior to the first dose of study drug.
14. Concurrent cytoreductive chemotherapy except hydroxyurea.
15. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to Tretinoin, Retinoids, soya, peanuts or Tranylcypromine.
16. Patients with psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
17. Patients with known epilepsy or patients with known psychiatric affections (bipolar disorder, schizophrenia, suicidal patients)
18. Pregnant or lactating and actively breastfeeding patients
19. Patients who are indignant to comply with nutritional conditions (see Protocol)
20. Poorly adjusted diabetes mellitus
21. Patients with hereditary Galactose-Intolerance, Lactase-Intolerance or Glucose-Galactose-Malabsorption
22. Known drug or alcohol abuse
23. Phaeochromocytoma or carcinoid tumor
24. Known cerebral vascular disease or other malformation of vessels (e.g. aneurysma)
25. Diabetes insipidus
26. Patients taking any of the following prohibited medication due to interaction with a) tretinoin and b) TCP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of the cumulative response rate (CR,CRp, CRi, PR) | every 28 day cycle
  Disease status will be assessed by bone marrow analyses

SECONDARY OUTCOMES:
number of participants with adverse events as a measure of safety and tolerability | one year
overall survival | 2 years
treatment effects of promotor genes | 2 Years
  To assess the cumulative incidence and degree of histone methylation of promotor genes in AML blasts after treatment with Tretinoin and tranylcpromine

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Mueller-Tidow, Prof., Principal Investigator — Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Universitaetsklinikum Halle, Halle, Germany